CLINICAL TRIAL: NCT00494624
Title: Efficacy of Systemic Glucocorticoid in the Treatment of Wheezing in Children
Acronym: VINKU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VINKU
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Wheezing
Keywords: Wheezing; virus; child
MeSH Terms: conditions — Respiratory Sounds; Virus Diseases | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: prednisolone

SUMMARY:
We can not predict which wheezing child younger than 3 years of age benefits from systemic glucocorticoid and which one does not. It is not known whether the differences in the efficacy are related to the differences in viral etiology, atopy, immunogical maturity or age of the patient. The study aims to answer the following questions: 1. What is the viral etiology of acute childhood expiratory wheezing? 2. What is the efficacy of prednisolone in relation to age, atopy and viral etiology in acute childhood wheezing? 3. Does prednisolone treatment increase risk for secundary bacterial infection in acute childhood expiratory wheezing? 4. What is the significance of inflammatory markers in predicting the efficacy of systemic steroid or patient outcome in acute childhood expiratory wheezing? Study will follow randomized, double blind, placebo-controlled parallel design. Study will start in Septemper 2000 and will be performed at the Department of Pediatrics, Turku University Hospital, Turku Finland. The study population will be 300 hospitalized wheezing children aged 3 months - 15 years. Investigational drug will be prednisolone, first dose 2 mg/kg, then 2 mg/kg/d/3 (max. 60 mg/vrk) p.o. for 3 d and comparative drug will be placebo tablet similar to investigational drug with the equal dosage. The primary outcome will be the time until ready for discharge. The study will provide new and important information for the diagnostics, treatment, disease outcome and prevention of acute childhood expiratory wheezing.

DETAILED DESCRIPTION:
Introduction

Extensive surveys have shown that 6-20 % of children have acute expiratory wheezing (1, 2). The lifetime prevalence of wheezing among 12-14-year-old children in the Western countries is 8-19 % (3, 4). The clinical illness is called bronchiolitis when occuring for the first time in infants younger than 12 months (5). When occuring later or recurring, beside bronchiolitis a diagnosis of wheezy bronchitis has been used (6). In older children wheezy bronchitis cannot be distinguished from virus-induced-asthma. In many countries the first expiratory wheezing attack at the age of > 3 years is diagnosed as asthma. To some extent, bronchiolitis, wheezy bronchitis, and asthma are expressions of the same pathologic process and at present there are no rigid criteria to separate these three illnessess.

Acute bronchiolitis is most commonly caused by respiratory syncytial virus (RSV) and wheezy bronchitis by rhinovirus infections (6 - 8). Exacerbations of asthma are induced in 80-85% of the cases by viral respiratory infections in children, mostly rhinovirus infections (7, 9).

It is well established that systemic glucocorticoids are the cornerstone in the management of acute asthma (10). However, systemic glucocorticoids do not appear to be effective in bronchiolitis in young children (11). Despite the lack of evidence for efficacy, glucocorticoids are used up to 60 % of patients with RSV bronchiolitis (12).

The unfavourable effects of glucocorticoids during viral infections have received increasing attention. For example, steroids have been found to increase the risk of acute otitis media during rhinovirus infections in children (13). In adults glucocorticoids have increased the titers of rhinovirus and the shedding of the virus from the pharynx (14, 15). It may be possible that glucocorticoids increase the severity of some viral respiratory tract infections.

Today, we can not predict which wheezing child younger than 3 years of age benefits from systemic glucocorticoid and which one does not. It is not known whether the differences in the efficacy are related to the differences in viral etiology, atopy, immunogical maturity or age of the patient.

Main Questions

1. What is the viral etiology of acute childhood expiratory wheezing?
2. What is the efficacy of prednisolone in relation to age, atopy and viral etiology in acute childhood expiratory wheezing?
3. Does prednisolone treatment increase risk for secundary bacterial infection in acute childhood expiratory wheezing?
4. What is the significance of inflammatory markers in predicting the efficacy of systemic steroid or patient outcome in acute childhood expiratory wheezing?

Rationale

The study provides new and important information for the diagnostics, treatment, disease outcome and prevention of acute childhood expiratory wheezing.

Design and setting

Study follows randomized, double blind, placebo-controlled parallel design. Study will start in Septemper 2000 and continue until June 2002 (except June and July 2001). The study will be performed at the department of pediatrics, Turku University Central Hospital, Turku Finland.

Subjects

The study population will be 300 patients. To allow detection of a 18-h difference (half of the average duration of stay in our hospital) in the time until ready for discharge between the prednisolone-treated group and the placebo groups (with an estimated standard deviation of 24 h) and to maintain an alpha error of 0.05 and a beta error of 0.20, the required size of the sample is 27 children for each treatment group in RSV bronchiolitis (16). No estimate is available for rhinovirus group. If patients are separated to different groups according to e.g. age or viral infection, 108 patients are needed. On the other hand to get 31 patients with a viral infection (viral infection in 80 % of patients with expiratory wheezing, and sensitivity of methods 69 %), 49 children are needed in each treatment group (to assess different subgroups, 196 children) (9, 17). To take account the variations of epidemics, a total of 300 children will be recruited. The estimated time to get enough patients, which need hospitalization for expiratory wheezing, will be 2 years at the department of pediatrics, Turku University Central Hospital, Turku, Finland.

Inclusion criteria

* age 3 months to 16 years
* hospitalization for expiratory wheezing
* written informed consent from the parents

Exclusion criteria

* Any chronic disease (other than allergy or asthma), e.g. heart disease, immune deficiency, or diabetes
* varicella and exposure to varicella if not previously have had it
* Systemic glucocorticoid 4 weeks prios to the study
* Severe disease that needs treatment in the intensive care unit or oxygen saturation below 92% despite of additional oxygen and frequent salbutamol inhalations

Study drugs

Investigational drug

Prednisolone, first dose 2 mg/kg, then 2 mg/kg/d/3 (max. 60 mg/vrk) p.o. for 3 d (5 mg tabletti, Prednisolon ®, Leiras, Finland).

Comparative drug

Placebo tablet similar to investigational drug (tablet, Leiras) will be given with the equal dosage.

Addministration of the drug

Tablets will be cut in four pieces, which mixt into jelly ot yogurt. If the child vomits, the drug will be given again after 30 min. If the child still vomits, he or she will be given equal dose of methylprednisolone or physiologic saline i.v. or i.m. (62,5 mg/ml inject, Solomet®, Orion, Finland).

Randomization

The randomization will be performed by an independent person not participating in the study. According to the randomization, each volunteer will be allocated to one treatment. Individual number 01 onwards will be assigned.

Protocol

The study physician will inform the subject and his or her guardian about the study and gives the subject information (Appendix 1). Guardian's written informed concent (Appendix 2) will be obtained after he or she has got acquainted with the test procedure. The subject can withdraw the consent to the study at any time. Guardian will be asked to fill the modified ISAAC questionaire (Appendix 3). New patients will enter the study at 8-10 a.m. and p.m.

The study is outlined in the study flow sheet (Appendix 4). The study physician will examine the patients twice daily at 8-10 a.m. and p.m. during the hospitalization (Appendix 5). The patients will be hospitalized until he or she does not wheeze or have breathing difficulties. After the hospitalization the patients will fill symptom diary for 2 weeks (Appendix 6). Follow-up visit will be 2 weeks after the hospitalization and follow-up telephone contact will be 2 months after the hospitalization. If the patient had a first wheezing episode, he or she will be re-examined 12 months after the study and oscillometric examination will be performed (if older than 24 months).

Nasal swap virological studies will also be performed to 60 healthy control children at outpatient clinic or surgical department in the Turku University Central Hospital during the study period.

Methods

Nasopharyngeal swap samples for virologic studies will be collected with 3 sterile cotton swaps which are dipped through the nostrils against nasal mucosa. These samples will be placed in a separate viral transport medium tubes for antigen, culture and PCR analysis.

Virus culture (influenza A and B , adeno-, RS-, parainfluenza type 1, 2 and 3 virus) was done by using the Ohio strain of HeLa cells and human foreskin fibroplasts according to routine procedure. Viral antigens (influenza A and B , adeno-, RS-, parainfluenza type 1, 2 and 3 virus) were detected by time-resolved fluoroimmunoassay with monoclonal antibodies (17). Reverse transcription-PCR assays were used for detection of corona-, rhino-, entero-, RS-, influenza A and B as well as human metapneumovirus (hMPV). The details of methods have been discribed earlier (18, 19). Virus-specific serum antibody titers (Influenza A and B virus, adenovirus, parainfluenza type 1/3 and 2 virus, RSV, HHV-6 and enterovirus IgG as well as for enterovirus also IgM) were determined by enzyme immunoassay (EIA) using antigen-coated solid phase and horsedish peroxidase conjugated rabbit antihuman IgG (Dako, Glostrup, Denmark). Three fold increase in IgG antibody titers was considered positive except four fold increase in RSV IgG antibody titers. Enterovirus was also considered positive if virus specific IgM was positive.

The influenssa A ja B , adeno , parainfluenssa type 1 , 2 and 3 as well as respiratory synsytial virus (RSV) antigen and culture, and rhino-, entero- and coronavirus PCR will be performed in the Department of Virology, Turku university, Finland. Human metapneumovirus PCR will be performed in the Department of Virology, Erasmus Medical Center, Rotterdam, The Netherlands. RSV A and B as well as Influenza virus A and B PCR will be performed in the National Health Institute, Helsinki, Finland. Viral and bacteral (C. pneumoniae, M. pneumoniae , S. pneumoniae, H. influenzae ja M. catarrhalis) will be performed in the National Health Institute, Oulu, Finland (17).

Expiratory nitric oxide will collected bed side with a bag collection system (Siemens) and analysed within 72 h at the Department of Clinical Physiology, Turku University Central Hospital, Turku, Finland (20). Oscillometric studies will be performed at the Department of Paediatric Turku University Central Hospital, Turku, Finland. Nasal cytokine (IL-8 and RANTES) measurements will be performed in the Children's Hospital, University of Texas Medical Branch, Galveston, Texas, USA. Other laboratory tests will be performed in the Central Laboratory, Turku University Central Hospital, Turku, Finland.

Primary endpoint: Our primary endpoint will be the time until ready for discharge, which will be defined as a duration of respiratory symptoms score >3 during hospital stay. The respiratory symptoms score, which will be assessed every 12 h during hospitalization, will consist of the degree of dyspnea (0=none, 1=mild, 2=moderate, 3=severe), type of breathing (0=normal, 1=use of stomach muscles, 2=use of intercostal muscles, 3=nasal flaring), severity of auscultatory findings on wheezing (0=none, 1=expiratory, 2=inspiratory and expiratory, 3=audible without stethoscope), and assessment of expiratory:inspiratory time (0=1:2, 1=1:1, 2=2:1, 3=3:1). An estimation of 6 h will be used for the last 12 h period between hospital assessments, i.e. the period during which the patient became ready for discharge.

Secondary endpoints: Oxygen saturation during hospital stay, wheeze and cough during two weeks after discharge from the hospital (assessed each day as none, mild, moderate or severe), readmission to the out-patient clinic or hospital for recurrent wheezing during a two-month period after discharge and blood eosinophil counts at discharge and two weeks later.

Adverse events

All adverse events encountered during the study period will be reported on the case record forms. The subjects will be urged to report any adverse events immetiately after appearance. All adverse events will be grated on a scale form 1 to 3, where 1 = mild, 2 = moderate and 3 = severe. The investigator will also be requested to judge the causality of each adverse event to the treatment (1 = not related, 2 = possibly related and 3 = probably related). If serious adverse effects occurs the sponsor shall be notified within 24 h by telephone and subsequently in writing by the investigator. All serious adverse events must be reported to national regulatory authorities within 24 hours of occurence.

Amendment of protocol

A new approval by the ethics committee has to be obtained before execution of any prospective deviation from the signed protocol.

Subject recruitment and information

Before recruitement, the guardian will be informed about the aims, character and risks of the study using the information text in the Subject Information (Appendix 1). After the subject has had sufficient time to acquaint himself with the information text, the investigator seeks for his written consent (Appendix 2). The original signed consent form will be retained by investigator. The investigator is responsible for informing all study team members of sufficient details of the study and the methods to be applied.

Ethical aspects

This study follows the recommendations for biomedical research involving human subjects (current revision of the Declaration of Helsinki of the World Medical Assembly). Prior to initiation of the study, the protocol, the subject information and the informed consent form will be submitted to and approved by the ethics committee of Turku University Central Hospital.

Data management and statistical analysis

The data will be collected in statistical software and the results will be analysed using statistical tests appropriate for parallel design. All study correspondence, records and documents related to the conduct of the study and the distribution of the investigational drug (e.g. diskettes, case record forms, concent forms and other pertinent information) must be retained by the investigator for a period of at least 15 years.

References

1. Ruuskanen O, Ogra PL. Respiratory syncytial virus. Curr Probl Pediatr 1993;23:50-79.
2. Martinez FD, Wright AL, Taussig LM, Holmberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med 1995;332:133-8.
3. Habbick BF, Pizzichini MM, Taylor B, Rennie D, Senthilselvan A, Sears MR. Prevalence of asthma, rhinitis and eczema among children in 2 Canadian cities: the International Study of Asthma and Allergies in Childhood. CMAJ 1999;160:1824-8.
4. Hesselmar B, Aberg B, Eriksson B, Aberg N. Asthma in children: prevalence, treatment, and sensitization. Pediatr Allergy Immunol 2000;11:74-9.
5. McIntosh K. Bronchiolitis and asthma: possible common pathogenetic pathways. J Allergy Clin Immunol 1976;57:595-604.
6. Mertsola J, Ziegler T, Ruuskanen O, Vanto T, Koivikko A, Halonen P. Recurrent wheezy bronchitis and viral respiratory infections. Arch Dis Child 1991;66:124-9.
7. Rakes GP, Arruda E, Ingram JM, et al. Rhinovirus and respiratory syncytial virus in wheezing children requiring emergency care. IgE and eosinophil analyses. Am J Respir Crit Care Med 1999;159:785-90.
8. Glezen PW, Greenberg SB, Atmar RL, Piedra PA, Couch RB. Impact of respiratory virus infections on persons with chronic underlying conditions. JAMA 2000;283:499-505.
9. Johnston SL, Pattemore PK, Sanderson G, et al. Community study of the role of viral infections in exacerbations of asthma in 9-11 year old children. BMJ 1995;310:1225-9.
10. Storr J, Barrell E, Barry W, Lenney W, Hatcher G. Effect of a single oral dose of prednisolonee in acute childhood asthma. Lancet 1987;1:879-82.
11. Roosevelt G, Sheehan K, Grupp Phelan J, Tanz RR, Listernick R. Dexamethasone in bronchiolitis: a randomised controlled trial. Lancet 1996;348:292-5.
12. Wang EEL, Law BJ, Boucher FD, et al. Pediatric investigators collaborative network on infections in Canada (PICNIC) study of admission and management variation in patients hospitalized with respiratory syncytial viral lower respiratory tract infection. J Pediatr 1996;129:390-5.
13. Ruohola A, Heikkinen T, Waris M, Puhakka T, Ruuskanen O. Intranasal fluticasone propionate does not prevent acute otitis media during viral upper respiratory infection in children. J Allergy Clin Immunol 2000;106:467-71.
14. Gustafson LM, Proud D, Hendley JO, Hayden FG, Gwaltney JM Jr. Oral prednisone therapy in experimental rhinovirus infections. J Allergy Clin Immunol 1996;97:1009-14.
15. Puhakka T, Mäkelä MJ, Malmström K, et al. The common cold: effects of intranasal fluticasone propionate treatment. J Allergy Clin Immunol 1998;101:726-31.
16. De Boeck K, Van der Aa N, Van Lierde S, Corbeel L, Eeckels R. Respiratory syncytial virus bronchiolitis: a double-blind dexamethasone efficacy study. J Pediatr 1997;131:919-21.
17. Mäkelä MJ, Puhakka T, Ruuskanen O, Leinonen M, Saikku P, Kimpimäki M, et al. Viruses and bacteria in the etiology of the common cold. J Clin Microbiol 1998; 36: 539 42.
18. Halonen P, Rocha E, Hierholzer J, Holloway B, Hyypiä T, Hurskainen P, Pallansch M. Detection of enteroviruses and rhinoviruses in clinical specimens by PCR and liquid-phase hybridization. J Clin Microbiology 1995;33:648-53.
19. van den Hoogen BG, de Jong JC, Groen J, Kuiken T, de Groot R, Fouchier RA, Osterhaus AD. A newly discovered human pneumovirus isolated from young children with respiratory tract disease. Nat Med 2001;7:719-24.
20. American Thoracic Society. Recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide in adults and children - 1999. Am J Respir Crit Care Med 1999; 160: 2104-17.

ELIGIBILITY:
Inclusion Criteria:

* age 3 months to 16 years
* hospitalization for expiratory wheezing
* written informed consent from the parents

Exclusion Criteria:

* Any chronic disease (other than allergy or asthma), e.g. heart disease, immune deficiency, or diabetes
* varicella and exposure to varicella if not previously have had it
* Systemic glucocorticoid 4 weeks prios to the study
* Severe disease that needs treatment in the intensive care unit or oxygen saturation below 92% despite of additional oxygen and frequent salbutamol inhalations

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2000-09; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
The time until ready for discharge

SECONDARY OUTCOMES:
Oxygen saturation during hospital stay
Wheeze and cough during two weeks after discharge from the hospital
Readmission to the out-patient clinic or hospital for recurrent wheezing during a two-month period after discharge
Blood eosinophil counts at discharge and two weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Jartti, MD, Principal Investigator — Turku University Hospital; Olli Ruuskanen, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Forsstrom V, Toivonen L, Homil K, Waris M, Pedersen CT, Bonnelykke K, Jartti T, Peltola V. Association of Asthma Risk Alleles With Acute Respiratory Tract Infections and Wheezing Illnesses in Young Children. J Infect Dis. 2023 Oct 18;228(8):990-998. doi: 10.1093/infdis/jiad075. PMID 36967681
- [Derived] Hurme P, Homil K, Lehtinen P, Turunen R, Vahlberg T, Vuorinen T, Camargo CA Jr, Gern JE, Jartti T. Efficacy of inhaled salbutamol with and without prednisolone for first acute rhinovirus-induced wheezing episode. Clin Exp Allergy. 2021 Sep;51(9):1121-1132. doi: 10.1111/cea.13960. Epub 2021 Jun 19. PMID 34062027
- [Derived] Lukkarinen M, Koistinen A, Turunen R, Lehtinen P, Vuorinen T, Jartti T. Rhinovirus-induced first wheezing episode predicts atopic but not nonatopic asthma at school age. J Allergy Clin Immunol. 2017 Oct;140(4):988-995. doi: 10.1016/j.jaci.2016.12.991. Epub 2017 Mar 25. PMID 28347734
- [Derived] Lukkarinen M, Lukkarinen H, Lehtinen P, Vuorinen T, Ruuskanen O, Jartti T. Prednisolone reduces recurrent wheezing after first rhinovirus wheeze: a 7-year follow-up. Pediatr Allergy Immunol. 2013 May;24(3):237-43. doi: 10.1111/pai.12046. Epub 2013 Feb 3. PMID 23373881